CLINICAL TRIAL: NCT00949260
Title: Hemodynamic Assessment of Healthy and Hypertensive Pregnant Women by Non-invasive Bio-reactance
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Other Study IDs: 09-01
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: PIH; pregnancy induced hypertension; pregnancy; bioimpedance; noninvasive monitoring; Cardiac Output; Blood Pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal, Non-Pregnant: Normal, non-pregnant patients will have 15 minutes of monitoring at rest, followed by a passive leg raising test.
- Normal, Pregnant: Normal, pregnant patients in their 3rd trimester will have 15 minutes of monitoring at rest, followed by a passive leg raising test.
- Pregnant, PIH: Pregnant patients in their 3rd trimester with pregnancy-induced hypertension that has not been treated will have 15 minutes of monitoring at rest, followed by a passive leg raising test.

SUMMARY:
The purpose of this study is to determine whether a noninvasive method of measuring certain aspects of blood circulation (e.g., blood pressure, cardiac output) is an accurate and reliable method to detect changes in pregnant patients. Specifically,the investigators are interested in patients diagnosed with high blood pressure during their pregnancy, as compared with normal pregnant patients. A noninvasive, accurate method of taking these measurements in pregnant patients is not currently available.

DETAILED DESCRIPTION:
During pregnancy, many aspects of blood circulation, such as blood pressure, heart rate, cardiac output, and stroke volume, adapt to accommodate the increasing needs of a pregnant body. The circulatory system works harder to provide blood flow to the placenta and the growing fetus.

Currently, the devices that can give physicians detailed information on the status of the blood circulation of normal patients and those with high blood pressure during pregnancy are invasive to varying degrees. However, recently, a new noninvasive hemodynamic monitor (NonInvasive Cardiac Output Monitoring: NICOM) was introduced to the market. In studies with non-pregnant patients, the NICOM has been found to be accurate, precise and reliable. However, it has yet to be studied in the field of Obstetrics.

The purpose of this study is to find out if the NICOM is an effective tool for monitoring hemodynamic changes in pregnant women, both with normal and high blood pressure. We are planning to compare the hemodynamic profiles of normal pregnant patients, hypertensive pregnant patients, and non pregnant patients as a control group. If this monitor proves to be reliable in assessing these changes in the pregnant patients, this could have a great impact in optimizing the care of the patients with different medical conditions in pregnancy, such as increased blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* PIH diagnosed in 3rd trimester, not yet treated
* healthy pregnant patients in 3rd trimester
* healthy non-pregnant women

Exclusion Criteria:

* under age 18 or above age 40
* refusal to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Our study population includes healthy non-pregnant and pregnant patients in their 3rd trimester, as well as pregnant patients in their 3rd trimester with pregnancy-induced hypertension (PIH). Both normal groups will be recruited from the outpatient day-unit (healthy volunteers). Patients with PIH may be sent to labour and delivery for monitoring by their obstetricians.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Index (CI) | 20 minutes

SECONDARY OUTCOMES:
Cardiac Output (CO) | 20 minutes
Blood Pressure (BP) | 20 minutes
Systemic Vascular Resistance (SVR) | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada